CLINICAL TRIAL: NCT03072303
Title: Pregnancy in Osteogenesis Imperfecta (OI) Registry
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: BBD7705; U01TR001263 (NIH)
Record Dates: First submitted 2017-01-25; First posted 2017-03-07 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Osteogenesis Imperfecta; Brittle Bone Disorders
Keywords: Brittle Bone; Osteogenesis Imperfecta; BBD; OI; Congenital Abnormalities; Congenital Bone Disorder; Lobstein Syndrome
MeSH Terms: conditions — Osteogenesis Imperfecta; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Web-based Survey — Patients will be sent an email invitation describing the study. If the participant wants to participate and is eligible, she will follow the survey link in the email message, which directs her to an IRB-approved online consent form. A unique survey link will be generated for each participant and included in the survey invitation, which is a customized email message. This link will allow the investigators to determine who completed the survey. The investigators will send repeat email invitations every two months (total of 3 invitations) to those invitees who have not yet participated. The investigators will allow approximately 6 months for enrollment and survey completion and expect that the study will close soon thereafter.

SUMMARY:
The purpose of this study is to learn about pregnancy outcomes in osteogenesis imperfecta (OI). Patients enrolled in the Brittle Bone Disorders (BBD) Contact Registry (CR) will be invited via email to participate in this study.

DETAILED DESCRIPTION:
Population: The RDCRN BBD Contact Registry helps researchers identify and recruit patients who are eligible for participation in future research studies. People eligible for enrollment in the RDCRN BBD Contact Registry include patients and parents of patients with Brittle Bone Disorders. All patients with BBD from the United States and around the world are encouraged to join.

Survey Administration: The investigators will administer a review of pregnancy outcomes survey and delineate the outcomes in pregnancies complicated by varying forms of OI. Patients will be sent an email invitation describing the study. If the participant wants to participate and is eligible, she will follow the survey link in the email message, which directs her to an IRB-approved online consent form. A unique survey link will be generated for each participant and included in the survey invitation, which is a customized email message. This link will allow the investigators to determine who completed the survey. The investigators will send repeat email invitations every two months (total of 3 invitations) to those invitees who have not yet participated. The investigators will allow approximately 6 months for enrollment and survey completion and expect that the study will close soon thereafter.

Data: The survey data will be collected and stored at the Rare Diseases Clinical Research Network's Data Management and Coordinating Center (DMCC) at the University of South Florida. All data collected will be sent to the database of Genotypes and Phenotypes (dbGaP) to be stored indefinitely.

ELIGIBILITY:
Inclusion Criteria:

* Female with OI who has delivered an infant of at least 24 weeks' gestation
* Participant in the BBD Contact Registry

Exclusion Criteria:

* Inability to provide informed consent and complete survey
* Males
* Women with OI who have not delivered children and gestations associated with higher order multiples

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The RDCRN BBD Contact Registry helps researchers identify and recruit patients who are eligible for participation in future research studies. People eligible for enrollment in the RDCRN BBD Contact Registry include patients and parents of patients with Brittle Bone Disorders. All patients with BBD from the United States and around the world are encouraged to join.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2019-03-13 (Actual); Study Completion 2019-09-13 (Actual)

PRIMARY OUTCOMES:
Pregnancy in OI Assessment | 1 year
  The goal of this survey is to characterize the course and outcome of pregnancy in individuals with OI. This is a self-report survey that will review pregnancy outcomes (maternal and fetal). Measures of pregnancy outcome will include 1) length of gestation, 2) mode of delivery, 3) neonatal outcomes including birth weight and length, 4) history of back pain or hip pain and or fractures during pregnancy or postpartum 5) number of maternal hospital admissions 6) calcium and vitamin D intake, 7) neonatal complications and 8) OI status in the fetus. One survey will be completed for each gestation (pregnancy).

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Krischer, Ph.D., Principal Investigator — University of South Florida; Deborah Krakow, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- RDCRN Data Management and Coordinating Center, University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McAllion SJ, Paterson CR. Musculo-skeletal problems associated with pregnancy in women with osteogenesis imperfecta. J Obstet Gynaecol. 2002 Mar;22(2):169-72. doi: 10.1080/01443610120113328. PMID 12521699
- [Background] Pennick V, Liddle SD. Interventions for preventing and treating pelvic and back pain in pregnancy. Cochrane Database Syst Rev. 2013 Aug 1;(8):CD001139. doi: 10.1002/14651858.CD001139.pub3. PMID 23904227
- [Background] Khovidhunkit W, Epstein S. Osteoporosis in pregnancy. Osteoporos Int. 1996;6(5):345-54. doi: 10.1007/BF01623007. PMID 8931028
- [Background] Pabinger C, Heu C, Frohner A, Dimai HP. Pregnancy- and lactation-associated transient osteoporosis of both hips in a 32 year old patient with osteogenesis imperfecta. Bone. 2012 Jul;51(1):142-4. doi: 10.1016/j.bone.2012.04.013. Epub 2012 May 3. PMID 22579778
- [Background] Choe EY, Song JE, Park KH, Seok H, Lee EJ, Lim SK, Rhee Y. Effect of teriparatide on pregnancy and lactation-associated osteoporosis with multiple vertebral fractures. J Bone Miner Metab. 2012 Sep;30(5):596-601. doi: 10.1007/s00774-011-0334-0. Epub 2011 Nov 23. PMID 22105654
- [Background] Moyer VA; U.S. Preventive Services Task Force. Screening for gestational diabetes mellitus: U.S. Preventive Services Task Force recommendation statement. Ann Intern Med. 2014 Mar 18;160(6):414-20. doi: 10.7326/M13-2905. PMID 24424622
- [Background] Hypertension in pregnancy. Report of the American College of Obstetricians and Gynecologists' Task Force on Hypertension in Pregnancy. Obstet Gynecol. 2013 Nov;122(5):1122-1131. doi: 10.1097/01.AOG.0000437382.03963.88. No abstract available. PMID 24150027
- [Background] Gaynes BN, Gavin N, Meltzer-Brody S, Lohr KN, Swinson T, Gartlehner G, Brody S, Miller WC. Perinatal depression: prevalence, screening accuracy, and screening outcomes. Evid Rep Technol Assess (Summ). 2005 Feb;(119):1-8. doi: 10.1037/e439372005-001. No abstract available. PMID 15760246
- [Background] National Vital Statistics Reports. Center for Disease Control. Volume 64, Number 1. (2015).
- [Background] Mercer BM. Preterm premature rupture of the membranes: current approaches to evaluation and management. Obstet Gynecol Clin North Am. 2005 Sep;32(3):411-28. doi: 10.1016/j.ogc.2005.03.003. PMID 16125041
- [Background] Callaghan WM, Kuklina EV, Berg CJ. Trends in postpartum hemorrhage: United States, 1994-2006. Am J Obstet Gynecol. 2010 Apr;202(4):353.e1-6. doi: 10.1016/j.ajog.2010.01.011. PMID 20350642
- [Background] Osterman MJ, Martin JA. Epidural and spinal anesthesia use during labor: 27-state reporting area, 2008. Natl Vital Stat Rep. 2011 Apr 6;59(5):1-13, 16. PMID 21553556
- [Background] Osterman MJ, Martin JA, Mathews TJ, Hamilton BE. Expanded data from the new birth certificate, 2008. Natl Vital Stat Rep. 2011 Jul 27;59(7):1-28. PMID 21848043
- [Background] Centers for Disease Control and Prevention (CDC). Update on overall prevalence of major birth defects--Atlanta, Georgia, 1978-2005. MMWR Morb Mortal Wkly Rep. 2008 Jan 11;57(1):1-5. PMID 18185492
- [Background] Wilcox AJ, Weinberg CR, O'Connor JF, Baird DD, Schlatterer JP, Canfield RE, Armstrong EG, Nisula BC. Incidence of early loss of pregnancy. N Engl J Med. 1988 Jul 28;319(4):189-94. doi: 10.1056/NEJM198807283190401. PMID 3393170
- [Background] Jones RK, Jerman J. Abortion incidence and service availability in the United States, 2011. Perspect Sex Reprod Health. 2014 Mar;46(1):3-14. doi: 10.1363/46e0414. Epub 2014 Feb 3. PMID 24494995
- [Background] Ory SJ. The national epidemic of multiple pregnancy and the contribution of assisted reproductive technology. Fertil Steril. 2013 Oct;100(4):929-30. doi: 10.1016/j.fertnstert.2013.06.004. Epub 2013 Jul 19. No abstract available. PMID 23876531
- [Background] Jebeile, H et al. A systematic review and meta-analysis of energy intake and weight gain in pregnancy. Institute of Medicine, Food and Nutrition Board, Committee on Nutritional Status During Pregnancy, part I: Nutritional Status and Weight Gain. National Academy Press, Washington, DC 2000. Am J Obstet Gynecol 12(2015).
- [Background] Zhang J, Savitz DA. Exercise during pregnancy among US women. Ann Epidemiol. 1996 Jan;6(1):53-9. doi: 10.1016/1047-2797(95)00093-3. PMID 8680626
- [Background] Wang SM, Dezinno P, Maranets I, Berman MR, Caldwell-Andrews AA, Kain ZN. Low back pain during pregnancy: prevalence, risk factors, and outcomes. Obstet Gynecol. 2004 Jul;104(1):65-70. doi: 10.1097/01.AOG.0000129403.54061.0e. PMID 15229002
- [Background] Mitchell AA, Gilboa SM, Werler MM, Kelley KE, Louik C, Hernandez-Diaz S; National Birth Defects Prevention Study. Medication use during pregnancy, with particular focus on prescription drugs: 1976-2008. Am J Obstet Gynecol. 2011 Jul;205(1):51.e1-8. doi: 10.1016/j.ajog.2011.02.029. Epub 2011 Apr 22. PMID 21514558